CLINICAL TRIAL: NCT07033754
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical Study to Assess the Effect of ProGenr8™ (Probiotic Supplement) on Immune Health in Teachers Prone to Upper Respiratory Tract Infection (URTI)
Brief Title: A Study to Assess the Effect Probiotic Supplement on Immune Health in Teachers Prone to Upper Respiratory Tract Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SB/240701/IP/URTI
Record Dates: First submitted 2025-03-06; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: URTI - Viral Upper Respiratory Tract Infection
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propionibacterium freudenreichii P.UF1 (Active Comparator): one capsule once a day with/beforebreakfast for 120 days
  Interventions: Dietary Supplement: Propionibacterium freudenreichii P.UF1
- Microcrystalline cellulose, calciumcarbonate, Mg Stearate, Sylysia (Placebo Comparator): one capsule once a day with/beforebreakfast for 120 days
  Interventions: Dietary Supplement: Microcrystalline cellulose, calciumcarbonate, Mg Stearate, Sylysia

INTERVENTIONS:
Dietary Supplement: Propionibacterium freudenreichii P.UF1 — one capsule once a day with/beforebreakfast for 120 days
  Arms: Propionibacterium freudenreichii P.UF1
Dietary Supplement: Microcrystalline cellulose, calciumcarbonate, Mg Stearate, Sylysia — one capsule once a day with/beforebreakfast for 120 days
  Arms: Microcrystalline cellulose, calciumcarbonate, Mg Stearate, Sylysia

SUMMARY:
The present study is a randomized, placebo-controlled, double-blind, parallel-group clinical studydesigned to assess the effects of IP on immune health in teachers prone to URTI. Approximately 179individuals aged between 18 and 50 years will be screened. Considering a screen failure of 20%,approximately 144 individuals will be randomized in a ratio of 1:1 to receive either the active orplacebo. The study will have at least 100 completed participants i.e. 50 participants in each studyarm after accounting for a dropout/withdrawal rate of 30% at the end of the study. The interventionand follow-up duration for all the study participants will be 120 days.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ready to give voluntary, written informed consent to participate in thestudy.
2. Male and female teachers aged between 18 to 50 years' (both values included) withmoderate physical activity level as per International Physical Activity Questionnaire -Short Form (IPAQ - SF).
3. Individuals with body mass index (BMI) between 22 kg per m2 to 32.0 kg per m2
4. High susceptibility to URTIs at least once every three months for last 1 year (at least 4to 6 episodes in a year).
5. Individuals who have active URTI episode at screening defined as "those having a scoreof less than equal to 5 for at least 2 symptoms out of runny nose, plugged nose,sneezing, sore throat, scratchy throat, cough or head congestion on the WURSS-21".
6. Commitment to adhere to routine diet and physical activity.
7. Willing to discontinue any immune-enhancing dietary supplements (e.g., prebiotics andfiber supplements, probiotics, Echinacea, fish oil, vitamin E, etc.) at least 1 one monthprior to screening.
8. Willing to discontinue sleep medications at least 1 month prior to screening and duringthe entire study duration.
9. Individuals willing to complete all study-related and clinical study visits as per theprotocol.

Exclusion Criteria:

1. Individuals with a history of rhinitis medicamentosa, anatomical nasal obstruction ordeformity, nasal reconstructive surgery, etc
2. Individuals taking prebiotics, probiotics, synbiotics or post-biotics supplements 1 monthprior to screening.
3. Individuals with known sensitivity to the investigational products or any excipients ofthe product.
4. Individuals with any clinically significant abnormalities of the upper respiratory tract(such as stridor, laryngomalacia, etc.).
5. Individuals suffering from lower respiratory tract infection (LRTI) of any origin.
6. Any individual not willing to follow the abstinence from any home-based remedies for common cold such as steam inhalation, decoctions, and vapor rub, etc.
7. Individuals with uncontrolled type 2 diabetes as assessed by fasting blood glucose lessthan equal to 126 mg per dL.
8. Individuals with uncontrolled hypertension on medication and with systolic bloodpressure less than 140 and or diastolic blood pressure less than equal to 90 mmHg.
9. Individuals who are unable to abstain from herbal or dietary supplements for URTI throughout the study period.
10. Vaccination against influenza or swine flu within 90 days prior to screening.
11. Those who have taken or should be taking or are taking antibiotics, antivirals, steroids,nasal decongestants, antihistamines, NSAIDs, or other medications that are expected to alleviate cold symptoms within two weeks prior to screening.
12. History of any significant neurological and psychiatric condition which may affect theparticipation and inference of the study's end points.
13. Participation in other clinical trials in last 90 days prior to screening
14. Individuals with substance abuse problems (within 2 years) defined as: a) Use ofrecreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine, tobaccoor smoking dependence. b) High-risk drinking as defined by consumption of 4 or morealcohol containing beverages on any day or 8 or more alcohol containing beverages perweek for women and 5 or more alcohol-containing beverages on any day or 15 or morealcohol containing beverages per week for men.
15. Individuals who have clinically significant following severe illness
16. Females who are pregnant/planning to be pregnant or lactating or taking any oralcontraceptives.
17. Any condition that could, in the opinion of the investigator, preclude the individual'sability to successfully and safely complete the study or that may confound studyoutcomes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
To Measure the effect of the 120 days' administration of IP on %population having one or more episodes of URTI during the study duration asassessed by Wisconsin Upper Respiratory Symptom Survey Questionnaire as compared to baseline and placebo. | Day 30,Day 90 & Day 120
  The WURSS-21 includes nine items assessing the impact of the URTI episode on an individual's quality of life i.e., the ability to think clearly, sleep well, breathe easily, exercise, work inside and outside the home, accomplish daily activities, interact with others and live one's personal life. All the items will be scored on an 8-point Likert scale ranging from 0 which depicts "absent or no impairment" to 1 (very mild), 3 (mild) 5(moderate), and 7 (severe). Participants will be instructed to fill this questionnaire whenever they have a URTI episode on all days throughout the study. An average of all WURSS-21 QoL scores will be calculated for every episode and considered to analyze the change in QoL as compared to baseline and placebo.

SECONDARY OUTCOMES:
To Measure the effect of IP in comparison to baseline and placebo on-Severity of the URTI episodes as assessed by Wisconsin Upper Respiratory Symptom Survey Questionnaire(WURSS-21) | From Date of Randomization upto 120 days
  In WURSS-21 All the items will be scored on an 8-point Likert scale ranging from 0, which depicts "absent or no impairment", to 1 (very mild), 3 (mild), 5 (moderate), and 7 (severe).43 The global score of WURSS-21 (question no. 1-19) ranges from 0-133 per day. Higher scores represent higher severity
To Measure the effect of IP in comparison to baseline and placebo on-Severity of the URTI episodes as assessed by Number of URTI episodes | From Date of Randomization upto 120 days
  the number of URTI episodes (frequency) and proves to be beneficial in individuals suffering from frequent URTI episodes
To Measure the effect of IP in comparison to baseline and placebo on -Body composition (Fat tissue, lean mass, fat free mass) as assessedby Dual Energy X-ray Absorptiometry -Gut microbiome analysis as assessed by Next Generation Sequencing | Day 0 and Day 120
  Dual Energy X-ray Absorptiometry Scans can assess fat content and total body composition with a high degree of precision that is comparable to hydrostatic weighing The investigation of the gut microbiota in a culture-independent manner has been made possible by next-generation sequencing technology, which has provided insights into the intricate and little-understood interactions between the gut microbiome and its host

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Nand Hospital, Vadodara, Gujarat
  - Lifeline Clinicand Diagnostics, Nashik, Maharashtra
  - AMF MorayaMultispecialityHospital, Pune, Maharashtra
  - ENT and VertigoClinic, Pune, Maharashtra
  - Madhumeh Clinic, New Delhi, National Capital Territory of Delhi
  - Janta Hospital &MaternityCentre, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No